CLINICAL TRIAL: NCT01996774
Title: Immunologic Profile of Children and Teenagers With Severe Allergy to Peanuts and Nuts After Induction of Tolerance: a Pilot Project
Brief Title: Immunologic Profile of Children With Severe Allergies to Peanuts and Nuts After Induction of Tolerance
Acronym: TOY
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P0013
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Immune Tolerance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood, serum, saliva

GROUPS / COHORTS (3):
- Child, peanut/ nut allergy, no treatment
- Child, peanut/nut allergy, tolerance
- Non allergic child, without atopia

SUMMARY:
Many authors propose the strict avoidance of allergenic food as the only treatment for children known to be allergic to certain food. However, it has been observed an increase of the frequency and severity of the allergic accidents in these children in the long term. Other teams have suggested treating these allergies (in particular peanut allergies) by controlled and progressive reintroduction of the allergenic food. A good tolerance and a prevention of allergic reactions consecutive to the ingestion of the same allergenic food were observed. The immunological mechanisms of this type of treatment are not well known.

A decrease of specific IgE and an increase of IgG4 have been observed in the case of egg allergies after this kind of treatment. Certain experiments realized in mice models testing the allergenic stimulation challenge showed an increase of lymphocytes T regulators (foxp3+ , CD4+, CD25+), stimulated by dendritic cells, and also an increase of interleukin 10, leading to the modification of the balance between Th1 and Th2.Our hypothesis is that after treating allergies by the reintroduction of the allergenic food, the immunological mechanism of acquisition of tolerance is associated to variations in populations of lymphocytes and in the activation or decrease of pro and anti-inflammatory cytokines. This reaction will be studied in two groups: 1. Children with a confirmed allergy to peanuts or nuts and 2. Children without antecedents of allergy or familiar atopy.

ELIGIBILITY:
Group 1:

Inclusion Criteria:

* Children (between 1 and 16 years old)known to have an allergy to peanuts and nuts detected by specific IgE, specific recombinant rArah (1 to 8) and R Cora and other allergens with a value superior or equal to 5KU/L.
* Child, parents or legal representatives have given informed consent to participate in the study after being informed in details about the protocol.

Exclusion Criteria:

* Immunodeficiency,
* Children or parents in disagreement with the study
* Children without standard diagnostic test at recruitment (oral provocation test vs. placebo)
* Children who reacted to placebo
* Children with uncontrolled asthma or respiratory disease
* Treatment with oral antihistaminic or corticoids one week before
* Neither Healthcare coverage nor insurance

Group 2:

Inclusion criteria

* Children (between 1 and 16 years old)known to have an allergy to peanuts and nuts detected by specific IgE, specific recombinant rArah (1 to 8) and R Cora and other allergens with a value superior or equal to 5KU/L
* Doubling the values of the threshold after second oral challenge compared to the tests of reference
* Child, parents or legal representatives have given informed consent to participate in the study after being informed in details about the protocol.

Exclusion Criteria:

* Immunodeficiency,
* Children or parents in disagreement with the study
* Children without standard diagnostic test at recruitment (oral provocation test vs placebo)
* Children who reacted to placebo
* Children with uncontrolled asthma or respiratory disease
* Treatment with oral antihistaminic or corticoids one week before
* Neither Healthcare coverage nor insurance

Group 3:

Inclusion criteria:

* Children (between 1 and 16 years old)
* No allergy to peanuts or nuts
* No antecedents of atopia
* Child, parents or legal representatives have given informed consent to participate in the study after being informed in details about the protocol

Exclusion Criteria:

* Immunodeficiency,
* Children or parents in disagreement with the study
* Children without standard diagnostic test at recruitment (oral provocation test vs. placebo)
* Children who reacted to placebo
* Children with uncontrolled asthma or respiratory disease
* Treatment with oral antihistaminic or corticoids one week before
* Neither Healthcare coverage nor insurance

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with allergy to peanuts and nuts hospitalized for initial diagnosis or for treatment in the Allergology Center of GHICL.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2012-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Allergen-specific biomarkers in blood and saliva | within the 15 days of subject enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Catalina ILIESCU, MD, PhD, Principal Investigator — Direction de la Recherche Médicale, Groupement des Hôpitaux de l'Institut Catholique de Lille
Locations (1):
- Groupement des Hôpitaux de l'Institut Catholique de Lille, Lomme, Nord, France